CLINICAL TRIAL: NCT05522673
Title: [11C]-(R)-Rolipram to Measure cAMP Signaling Before and After Ketamine
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10000824; 000824-M
Record Dates: First submitted 2022-08-30; First posted 2022-08-31 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-01

CONDITIONS: Depression
Keywords: PET Imaging; Inflammation; Ketamine; Depression
MeSH Terms: conditions — Depression; Inflammation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects with major depression disorder (MDD) (Other): Participants with major depressive disorder received 20 mCi of [11C](R)-rolipram intravenously for two PET scans, prior to and after ketamine infusion as well as brain MRI
  Interventions: Drug: 11(R)-rolipram

INTERVENTIONS:
Drug: 11(R)-rolipram — Injected IV followed by PET scanning

SUMMARY:
Background:

Major depressive disorder (MDD) may have many underlying causes. One theory is that brain cells with low levels of a molecule called cyclic AMP (cAMP) may cause depression. A drug called ketamine may increase the levels of cAMP in a person's brain cells.

Objective:

To find out if administering ketamine to people with depression affects cAMP levels in their brains.

Eligibility:

People aged 18 to 70 with MDD who are enrolled in another NIH study that uses ketamine.

Design:

Participants will visit the NIH clinic 5 times in up to 6 weeks. Some of the visits may be spread out over more than 1 day.

Participants will be screened. They will have a physical exam with blood and urine tests. They will have a test of their heart function. They will have a psychiatric evaluation. They will answer questions about their family history and mental health.

Participants will have a positron emission tomography (PET) scan. A small amount of a radioactive drug will be injected into a vein in their arm. Participants will lie on a bed that slides in and out of a doughnut-shaped machine that records images of their brains. They will have their heads in a holder to prevent movement. Each scan will last up to 2 hours.

After their first PET scan, participants will receive ketamine in a different study they are enrolled in. Then they will come back for another PET scan with the radioactive drug.

Participants will also have another scan called an MRI. They will lie on a table that slides into a metal tube. They will lie still for up to an hour....

DETAILED DESCRIPTION:
Study Description:

This study will test the effects of ketamine infusion on the cAMP system in human brain to determine if ketamine mediates its antidepressant effects at least in part due to modulation of cAMP signaling.

Objectives:

Primary Objective: To determine if ketamine infusions in depression causes increases in cAMP signaling as measured by [11C](R)-rolipram binding.

Secondary Objectives: To determine if increases in [11C](R)-rolipram correlate with symptomatic improvement in major depressive symptoms.

Endpoints:

Primary Endpoint: measurement of PDE4 density (volume of distribution VT) in brains of individuals with major depressive disorder (MDD) before and after administration of ketamine.

Secondary Endpoints: Clinical rating scales of depression, including MADRS, HAM-D.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients:

In order to be eligible for this study, MDD participants must meet all of the following criteria:

1. Be male or female, aged 18 to 70 years old.
2. Female participants of childbearing potential must be using a medically acceptable means of contraception.
3. Participants must be in good general health as evidenced by medical history and physical examination.
4. Each participant must have a level of understanding sufficient to agree to all required tests and examinations and sign an informed consent document.
5. All participants must have undergone a screening assessment under protocol 01-M-0254, 'The Evaluation of Patients with Mood and Anxiety Disorders and Healthy Participants'.
6. Participants must be enrolled in the ketamine arms of protocols 19-M-0107 'Ketamine and AMPA', 17-M-0060 'Neuropharmacology of Ketamine', or 15-M-0188 'Neurobiology of Suicide'.
7. Participants must fulfill DSM-5 criteria for major depression (MDD) without psychotic features, as based on clinical assessment and structured diagnostic interview (SCID-P).
8. Participants must have an initial score on the MADRS >= 18 or HAM-D >= 15 within two weeks of study entry.
9. Participants with stable medical conditions as assessed by their primary care provider (PCP) and/or in-house clinician are permitted to join the study.
10. Patients must qualify for ketamine administration, usually defined as lack of response to two adequate lifetime antidepressant trials, with [at least] one in the current major depressive episode, operationally defined using the Antidepressant Treatment History Form (ATHF); a failed adequate trial of ECT [or TMS] would count as an adequate antidepressant trial.
11. Participants must have their radial artery pulse checked for the presence of adequate ulnar collateral flow and the absence of any metal or foreign objects in both wrists.
12. Participants must agree to adhere to the lifestyle considerations.

EXCLUSION CRITERIA:

Participants with MDD who meet any of the following criteria will be excluded from participation in this study:

1. Clinically significant abnormalities on EKG or laboratory testing. This includes CBC; acute care panel [Na, K, Cl, CO2, creatinine, glucose, urea nitrogen); hepatic panel (alkaline phosphatase, alanine transaminase (ALT), aspartate aminotransferase ([AST), bilirubin total, and bilirubin direct]; mineral panel (albumin, calcium, magnesium, phosphorus); glucose; prothrombin and partial prothrombin tests.
2. Current psychotic features, a diagnosis of schizophrenia or any other psychotic disorder as defined in the DSM-5.
3. Participants with a history of DSM-5 substance use disorder (except for caffeine or nicotine dependence) within the preceding three months. In addition, participants must not have substance use disorder or alcohol use disorder. However, alcohol or cannabis use by themselves are not exclusion criteria, unless that use affects the function of daily life.
4. Participants who, in the investigator s judgment, pose a current serious suicidal or homicidal risk.
5. Participants who have a history of aggressive behavior towards others.
6. Participants who have an unstable medical condition that, in the opinion of the investigators, makes participation unsafe (e.g., an active infection or untreated malignancy).
7. Are unable to travel to the NIH.
8. Have recent exposure to radiation related to research (e.g., PET from other research) that, when combined with this study, would be above the allowable limits.
9. Have an inability to lie flat and/or lie still on the camera bed for at least two hours, including claustrophobia, overweight greater than the maximum for the scanner, and uncontrollable behavioral symptoms, which will be screened by an interview with the participant during the screening visit.
10. Are unable to have an MRI scan (e.g., because of pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, shrapnel fragments, or metal fragments in the eye.
11. Be National Institute of Mental Health (NIMH) staff or an NIH employee who is a subordinate/relative/co-worker of the investigators.
12. Pregnancy
13. HIV infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000824-M.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With Major Depression Disorder (MDD): Participants with major depressive disorder received 20 mCi of [11C](R)-rolipram intravenously for two positron emission tomography (PET) scans, prior to and after ketamine infusion as well as brain MRI
Period: Overall Study
Arm/Group | Subjects With Major Depression Disorder (MDD)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects With Major Depression Disorder (MDD)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Whole Brain Total Distribution Volume (VT)
Description: Participants received 11C-R-Rolipram during PET scan and were scanned for 90 minutes with arterial blood sampling. Volume of distribution was calculated using two-tissue compartmental modeling. Participants had one PET scan pre-Ketamine and a second PET scan post-Ketamine administration.
Time Frame: 90 minutes after injection of 11C-R-Rolipram
Population: Analysis included participant who completed the study
Measure: Number; unit: mL x cm^3
Arm/Group | Subjects With Major Depression Disorder (MDD)
Number analyzed (Participants) | 1
mL x cm^3
  Pre-Ketamine | 0.512639
  Post-Ketamine | 0.443411

2. Secondary Outcome: Measure of Level of Depression Using Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: Participants rated level of depression using Montgomery-Åsberg Depression Rating Scale (MADRS). MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Each item yields a score of 0 to 6 with overall score ranging from 0 to 60. Higher MADRS score indicates more severe depression. Scores were measured at two visits, pre-Ketamine administration and a second visit post-Ketamine administration.
Time Frame: Within two weeks of start of study (Pre) and within 7 days of Ketamine infusion (Post)
Population: Analysis included participant who completed the study
Measure: Number; unit: score on a scale
Arm/Group | Subjects With Major Depression Disorder (MDD)
Number analyzed (Participants) | 1
score on a scale
  Pre-Ketamine | 28
  Post-Ketamine | 25

3. Secondary Outcome: Measure of Level of Depression Using the Hamilton Depression (HAM-D) Rating Scale
Description: Participants rated level of depression using the Hamilton Depression (HAM-D) Rating Scale. The HAM-D is a clinician-administered depression assessment scale which contains 17 items pertaining to symptoms of depression experienced over the past week. Eight items are rated 0-4 and nine items are rated 0-2 for a minimum score of zero and a maximum score of 50. Higher value indicates worsening depression. Scores were measured at two visits, prior to PET scan pre-Ketamine and a second visit post-Ketamine administration.
Time Frame: Within two weeks of start of study (Pre) and within 7 days of Ketamine infusion (Post)
Population: Analysis included participant who completed the study
Measure: Number; unit: score on a scale
Arm/Group | Subjects With Major Depression Disorder (MDD)
Number analyzed (Participants) | 1
score on a scale
  Pre-Ketamine | 17
  Post-Ketamine | 16

ADVERSE EVENTS:
Time Frame: Up to 24 hours for each visit for a total of two visits
Arm/Group | Subjects With Major Depression Disorder (MDD)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Study was prematurely terminated due to low recruitment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT05522673/Prot_SAP_000.pdf